CLINICAL TRIAL: NCT02770755
Title: Registry of Celution Device for the Processing of Adipose Derived Regenerative Cells (ADRCs) and Healing in Muscle and Ligament Sports Injuries (ACHILLES)
Brief Title: Registry of Celution Device for Processing ADRCs and Healing in Muscle and Ligament Sports Injuries
Acronym: ACHILLES
Status: Withdrawn | Type: Observational
Why Stopped: Corporate decision
Sponsor: Cytori Therapeutics (Industry)
Responsible Party: Sponsor
Other Study IDs: ACHILLES
Record Dates: First submitted 2016-03-15; First posted 2016-05-12 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Muscle Tear

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year

SUMMARY:
This registry study will compile information about patients who are scheduled to receive or have received Adipose Derived Regenerative cells (ADRCs) prepared by Celution device to treat muscle and ligament sports injuries.

ELIGIBILITY:
Inclusion Criteria:

* Males or females > 18 of age
* Patients with sports related muscle tear (≥5%) with or without ligament injury as confirmed by ultrasound or MRI with onset of injury in preceding year
* Pain in the affected area at rest and/or movement
* Weakness or inability to use affected muscle

Exclusion Criteria:

* Muscle tear <5% or unrepaired complete tears or ruptures on ultrasound or MRI
* Known spine or disc disease or symptomatic impingement of nerve root
* Known neuromuscular disease (e.g., amyotrophic lateral sclerosis, muscular dystrophy)
* History of documented nerve damage in the affected limb
* Tears involving open wounds
* Tears requiring surgical repair
* Pregnant or lactating status. Pregnancy as determined by a positive pregnancy test at screening or baseline

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are scheduled to receive or have received Adipose Derived Regenerative Cells (ADRCs) prepared by Celution device to treat muscle and ligament sports injuries.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Estimated); Study Completion 2017-05 (Estimated)

PRIMARY OUTCOMES:
Change in magnitude of muscle tear as assessed by ultrasound or MRI | 42 days

SECONDARY OUTCOMES:
Change in magnitude of muscle tear as assessed by ultrasound or MRI | 21 days
% of patients with complete healing as measured by ultrasound or MRI | Days 7, 14, 21, 42 and 90
Change in pain | Days 7, 14, 21, 42 and 90
  Change in pain assessed via patient questionnaires
Change in function | Days 7, 14, 21, 42 and 90
  Change in function assessed via patient questionnaires

OTHER OUTCOMES:
Recurrent muscle tears | Days 7, 14, 21, 42 and 90
  Number of recurrent muscle tears

CONTACTS AND LOCATIONS:
Overall Officials: Steven Kesten, M.D., Study Chair — Cytori Therapeutics
Locations (1):
- The Football Association, Wembley, United Kingdom